CLINICAL TRIAL: NCT01807897
Title: Oxygen Versus PAP for Treatment of Sleep Apnea in Chronic Heart Failure
Brief Title: Oxygen Versus PAP for Sleep Apnea in Heart Failure
Acronym: OPTIMAL-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLIN-008-12S
Record Dates: First submitted 2013-03-01; First posted 2013-03-08 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure; Sleep Apnea Syndromes
Keywords: Heart Failure; Sleep Apnea; Ventricular Ejection Fraction; Exercise Test
MeSH Terms: conditions — Heart Failure; Sleep Apnea Syndromes | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Continuous positive airway pressure (CPAP) and supplemental oxygen
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- CPAP (Experimental): Nocturnal continuous positive airway pressure
  Interventions: Device: Continuous positive airway pressure; Behavioral: Healthy Lifestyle and Sleep Education
- NSO (Experimental): Nocturnal supplemental oxygen
  Interventions: Device: Nocturnal supplemental oxygen; Behavioral: Healthy Lifestyle and Sleep Education
- HLSE (Other): Healthy lifestyle and sleep education control
  Interventions: Behavioral: Healthy Lifestyle and Sleep Education

INTERVENTIONS:
Device: Continuous positive airway pressure — Nocturnal continuous positive airway pressure, titrated to minimize apnea-hypopnea index
  Other Names: CPAP
  Arms: CPAP
Device: Nocturnal supplemental oxygen — Nocturnal supplemental oxygen, titrated to 2-4 liters/minute with target of eliminating nocturnal hypoxemia
  Other Names: NSO
  Arms: NSO
Behavioral: Healthy Lifestyle and Sleep Education — A 60-minute educational intervention with slide show and printed materials, educating the patient in healthy sleep habits and heart-healthy lifestyle
  Other Names: HLSE

SUMMARY:
The purpose of this study is to compare three treatment modalities for central, or mixed obstructive and central, sleep apnea in patients with chronic heart failure and reduced ejection fraction. The modalities to be tested are nocturnal supplemental oxygen (NSO) and continuous positive airway pressure (CPAP). The main outcome measures will be left ventricular ejection fraction on echocardiogram and peak oxygen consumption on cardiopulmonary exercise testing.

DETAILED DESCRIPTION:
Chronic heart failure (HF) is a highly prevalent disease, with a lifetime risk of approximately 20%. Sleep apnea is a common co-morbid condition, occurring in approximately half of patients with chronic HF, and often has predominantly central or mixed obstructive and central characteristics. Although it is associated with increased mortality in patients with HF, sleep apnea is usually asymptomatic and patients are therefore often unwilling to accept standard therapy with positive airway pressure. At the outset of this study, there were three treatment modalities currently recommended by the American Academy of Sleep Medicine for the treatment of predominantly central sleep apnea in HF patients: nocturnal supplemental oxygen (NSO), continuous positive airway pressure (CPAP) and adaptive servo-ventilation (ASV). Recently, ASV was found to increase mortality in patients with heart failure with reduced ejection fraction and central sleep apnea. There are only limited data on the comparative efficacy and tolerability of these three modalities. The present study is designed to compare these modalities with respect to effects on ventricular function, exercise capacity, and other measures of cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Veteran receiving care within the Veterans Health Administration healthcare system
* Age 18 years
* Physician diagnosis of chronic heart failure, American Heart Association Stage C-D
* LVEF <45%
* No change in active cardiac medications for 4 weeks prior to randomization
* Ability to provide informed consent
* Moderate to severe central or mixed central and obstructive sleep apnea, defined as an apnea-hypopnea index (AHI) 15 events per hour, with a central AHI >5 events/hour

Exclusion Criteria:

* Hospitalization for acute decompensated HF within previous 30 days
* Hospitalization for myocardial infarction or cardiac surgery within previous 90 days
* Presence of a left ventricular assist device
* History of heart transplantation
* Poorly controlled hypertension (>170/>110)
* Poorly controlled diabetes (HbA1c > 9.0)
* Severe renal failure with estimated glomerular filtration rate <30 ml/min
* Prior stroke with functional impairment or other severe, uncontrolled medical problems that may impair ability to participate in the study exams, based on medical history and review of medical records
* Severe chronic insomnia, with reported usual sleep duration <4 hours
* Severe daytime sleepiness, defined as Epworth Sleepiness Scale score 18 or higher or a report of falling asleep driving during the previous year, and deemed a safety risk by study physician
* Awake resting oxyhemoglobin saturation <89%
* Pregnancy
* Smoking by subject or other person in the subject's bedroom, or other open flame in bedroom
* Current use of a positive airway pressure device (including continuous or bi-level positive airway pressure or adaptive servo-ventilation) or supplemental oxygen therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Gottlieb, MD MPH, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxygen: Nocturnal supplemental oxygen
  Nocturnal supplemental oxygen: Nocturnal supplemental oxygen, titrated to 2-4 liters/minute with target of eliminating nocturnal hypoxemia
  Healthy Lifestyle and Sleep Education: A 60-minute educational intervention with slide show and printed materials, educating the patient in healthy sleep habits and heart-healthy lifestyle
Period: Overall Study
Arm/Group | CPAP | Oxygen | HLSE
Started | 31 | 29 | 14
Completed | 24 | 27 | 13
Not Completed | 7 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CPAP | Oxygen | HLSE | Total
Number analyzed (Participants) | 31 | 29 | 14 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 14
  >=65 years | 26 | 24 | 10 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (10.2) | 71.7 (8.3) | 70.5 (8.1) | 71.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 31 | 28 | 14 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 4
  Not Hispanic or Latino | 27 | 25 | 13 | 65
  Unknown or Not Reported | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 2 | 8
  White | 23 | 22 | 12 | 57
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 3 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction
Description: Standard transthoracic 2-dimensional and Doppler echocardiography will be performed. M-mode measurements of LV dimensions will be performed and analyzed according to the American Society of Echocardiography recommendations and LVEF measured using the modified Simpson's method. Measurement is change from baseline in LVEF.
Time Frame: 3 months
Population: All participants with both baseline and follow-up echocardiograms. There were 5 dropouts from the CPAP group, 2 from the NSO group and 1 from the HLSE group.
Measure: Mean (Standard Deviation); unit: percent of LV diastolic volume
Arm/Group | CPAP | Oxygen | HLSE
Number analyzed (Participants) | 24 | 27 | 13
percent of LV diastolic volume | 1.63 (4.88) | 1.69 (8.33) | 4.42 (4.85)

2. Secondary Outcome: Peak Oxygen Consumption (VO2 Peak)
Description: Treadmill exercise testing will be performed using a motor-driven treadmill and a modified Naughton protocol, with a lightweight disposable pneumotach device positioned in the participant's mouth interfaced with a metabolic cart. Change in VO2 peak between baseline and final visit will be the co-primary outcome of the study. Secondary outcome measures from cardiopulmonary exercise testing include VO2 at anaerobic threshold and VE/VCO2 slope.
Time Frame: 3 months
Population: All randomized participants completing baseline and follow-up cardiopulmonary exercise testing
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | CPAP | Oxygen | HLSE
Number analyzed (Participants) | 17 | 21 | 7
ml/kg/min | -0.40 (2.59) | 0.11 (4.75) | -1.54 (2.39)

3. Secondary Outcome: 24-hour Ambulatory Blood Pressure
Description: 24-hour blood pressure will be measured using a blood pressure cuff that is connected by rubber tubing to a small pressure monitoring device, programmed to measure BP at 20 minute intervals during the day and 30 minute intervals at night (11 PM to 7 AM) for a period of 24 hours. The investigators will assess 24-hour mean arterial pressure as the primary blood pressure outcome, with additional assessment of nocturnal versus diurnal blood pressure effects.
Time Frame: 3 months
Population: Participants completing 24-hour ambulatory BP monitoring at final visit
Measure: Mean (Standard Deviation); unit: torr
Arm/Group | CPAP | Oxygen | HLSE
Number analyzed (Participants) | 9 | 14 | 5
torr | 87.5 (8.5) | 88.0 (9.1) | 77.4 (9.9)

ADVERSE EVENTS:
Time Frame: 3 months
Description: AE data collected at 1, 2, 4, and 8 weeks of follow-up and at final visit.
Arm/Group | CPAP | Oxygen | HLSE
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/31 | 4/29 | 2/14
Other Adverse Events (participants affected / at risk) | 10/31 | 13/29 | 4/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (N=31) | Oxygen (N=29) | HLSE (N=14)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Heart failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) — Exacerbation of heart failure symptoms requiring hospitalization
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Fall with injury requiring hospitalization
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Atrial fibrillation requiring intervention
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalized for chest pain
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CPAP (N=31) | Oxygen (N=29) | HLSE (N=14)
Increased dyspnea (Cardiac disorders) | 5 (5) | 4 (4) | 2 (2) — Dyspnea new or worse shortness of breath since prior contact
Chest discomfort (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) — New or worse discomfort or pain in chest since prior contact
Excessive sleepiness (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0) — Sleepiness interfering with work or driving since prior contact
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Decreased renal function (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (General disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall with injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT01807897/Prot_SAP_000.pdf